CLINICAL TRIAL: NCT01918150
Title: A French, Multicentric, Randomized, Simple Blind, Superiority Study Comparing the Efficiency and the Safety at 24 Months of the Stent Titan2 Versus Bare Metal Stent in Cobalt-Chrome in All Comers Patients Among Which 40 % Present an ACS.
Brief Title: Comparative Phase IV Study: Efficacy And Safety of TiTAN2 Versus COBALT-CHROME Stents- EVIDENCEII
Acronym: EVIDENCE II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hexacath, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HXF-CT2-20111
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Silent Myocardial Infarction; Stable Angina; Acute Coronary Syndrome
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TITAN 2 stent - Hexacath France (Experimental): Patients receiving Titan 2 stents (percutaneous coronary intervention)
  Interventions: Device: Titan 2 stents
- Cobalt-Chromium BMS - Any firm (Active Comparator): Patients receiving Cobalt-Chromium Bare Metal Stents (free of any coating)(percutaneous coronary intervention)
  Interventions: Device: Cobalt-Chromium Bare Metal Stents

INTERVENTIONS:
Device: Titan 2 stents — The intervention is called Percutaneous Coronary Intervention (PCI); Commonly known as coronary angioplasty or simply angioplasty, it is a non-surgical procedure used to treat the stenotic (narrowed) coronary arteries of the heart found in coronary heart disease. PCI is usually performed by an interventional cardiologist.
  Arms: TITAN 2 stent - Hexacath France
Device: Cobalt-Chromium Bare Metal Stents — The intervention is called Percutaneous Coronary Intervention (PCI); Commonly known as coronary angioplasty or simply angioplasty, it is a non-surgical procedure used to treat the stenotic (narrowed) coronary arteries of the heart found in coronary heart disease. PCI is usually performed by an interventional cardiologist.
  Arms: Cobalt-Chromium BMS - Any firm

SUMMARY:
The purpose of this study is to compare the effectiveness and safety, at 24 months, of the TITAN2 stent to any bare-metal stent (BMS) in Cobalt-Chromium in a population presenting an indication for these stents among 40% of which present an acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
The EVIDENCE II trial is a post-registration study for TITAN2 stent initiated on the request of the French Health Authorities' (HAS) in June 2009 for the next renewal of registration on the list of reimbursable products and services in France.

The study is so designed to compare the effectiveness and safety at 24 months of the TiTAN2 versus Cobalt-Chromium BMS randomly assigned. As a part of the secondary objectives, a cost-effectiveness study is also planned.

The comparators are cobalt chromium stents CE marketed and free of any coating (nude BMS).

All will be used in their authorized indications.

A total of 1350 patients will be included over a period of a year or more and followed for 24 months for the primary endpoint (MACE rate at 24 months in the overall population : cumulative incidence of cardiac deaths, MI and target lesion revascularization (TLR)).

Patients will also be clinically followed at 6 and 12 months . Medico economic datas are to collect at a similar time point.

An independent Clinical Event Committee, unaware of the treatment allocation, will be in charge of the adjudication of all the cardiac events including MACE (main objective)collected.

The calculation of the number of subjects specifies that 1350 patients are needed to meet the primary endpoint of the study.

Enrolled patient will be randomly assigned in a 2:1 fashion as follows :

* 900 patients in TITAN2 arm including 360 with ACS (Arm A)
* 450 patients in Cobalt-chromium arm including 180 with ACS (Arm B) In case of more than one stent needed, the protocol mandated using the same stent than the one assigned in all the lesions treated.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic de novo coronary lesion involving one or two vessels
* Patient presenting a lesion with > 50% stenosis
* Patient who must undergo a percutaneous coronary intervention (PCI) in the indications of Cobalt-chromium bare metal stents and TITAN2 stents and being able to be indifferently treated with one or the other of these stents.
* Written informed consent
* Expected survival > 2 years
* Patient reachable by phone throughout the duration of the study.

Exclusion Criteria:

* Pregnant/Lactating women
* Women of childbearing potential (last menstrual period <12 months) not using effective contraception
* Patient under legal protection
* Indication of coronary artery bypass graft surgery (CABG)
* History of coronary artery bypass graft surgery (CABG)
* Intrastent restenosis lesion
* Bifurcation lesion with the exception of those treated with a standardized approach (provisional stenting with final kissing in the side branch)
* Left main coronary lesion
* Ostial target lesion
* Previous drug-eluting stenting
* Previous bare metal stenting or balloon angioplasty in the 12 months prior the inclusion; if this implantation involved the target artery, separate the new implanted stent at a distance ≥ 10 mm.
* History of stent thrombosis
* Heavily calcified lesion
* Use of the Rotablator
* Left ventricular ejection fraction (LVEF) < 30%
* Cardiac arrest, cardiogenic shock or severe heart failure (Killip stage III or IV)
* Severe chronic renal failure (creatinine clearance <30 ml min)
* Cardiac or renal transplantation
* Major surgery within the last 14 days
* Surgery scheduled within 30 days (non-ACS patients) or 12 months (if ACS) at the time of the randomization
* History of major bleeding
* Pathology with major risk of bleeding or any condition, allergy or intolerance which is incompatible with anticoagulation and / or extended antiplatelet therapy
* Known allergy to Titanium, Nickel, Cobalt or Chromium
* Patient currently participating in another clinical trial
* Non-compliant patient (treatment and follow-up)
* Patient living abroad

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
MACE | 24 months
  The primary endpoint (MACE) is the composite of cardiac death, (Myocardial Infarction) MI and target lesion revascularization (TLR).
  These events will be collected post-procedure during the patient's hospitalization and at 6 , 12 and 24 month follow-up.

SECONDARY OUTCOMES:
Medico economic evaluation | 24 months
  Data collection of acts and diagnosis specific codes related to any adverse event with hospitalization in relation with the endoprothesis allocated.
  It will be then analyzed by an dedicated expert who will be able to appreciate a cost/efficiency rate for each treatment arm.
Target Lesion Revascularization (TLR ) rate | 24 months
  Any study stent restenosis leading to a procedure or a surgery to treat it.
Stent thrombosis rate | 24 months
  Stent thrombosis will be evaluated as per the ARC classification (ie degree of evidence and time to event)
Success of the procedure | 24 months
  Defined as an efficient reintroduction of the blood flow in the target vessel post angioplasty.
  It's a "YES/NO" question.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RIOUFOL, Pr, Principal Investigator — Hospices Civils de Lyon- Bron - France
Locations (42):
- France (42):
  - Clinique Claude Bernard, Albi
  - Clinique de l'Europe, Amiens
  - Hôpital Sud, Amiens
  - CHU Angers, Angers
  - CH Henri Duffaut, Avignon
  - Clinique La Fourcade, Bayonne
  - Polyclinique de Bois Bernard, Bois-Bernard
  - CHU Côte de Nacre, Caen
  - CH Cannes, Cannes
  - Centre hospitalier Louis Pasteur, Chartres
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Albert Schweitzer, Colmar
  - Ch Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Laënnec, Creil
  - CHU de Grenoble, Grenoble
  - Groupe Hospitalier Mutualiste, Grenoble
  - Centre Hospitalier Général, Haguenau
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny
  - Centre Hospitalier de Lille, Lille
  - HCL Bron, Lyon
  - HCL Croix-Rousse, Lyon
  - Clinique Beauregard, Marseille
  - Hôpital Nord, Marseille
  - Clinique Les Fontaines, Melun
  - Hôpital Emile Muller, Mulhouse
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU Caremeau, Nîmes
  - Clinique Alleray Labrouste, Paris
  - HIA Val de Grâce, Paris
  - Hôpital Saint-Joseph, Paris
  - CH Pau, Pau
  - Clinique Saint-Martin, Pessac
  - Hôpital Claude Galien- ICPS, Quincy-sous-Sénart
  - Clinique Saint Laurent, Rennes
  - Clinique Saint-Hilaire, Rouen
  - CH Saint-Brieuc, Saint-Brieuc
  - CHI Toulon La Seyne, Toulon
  - Clinique Pasteur, Toulouse
  - Hôpital de Rangueil, Toulouse
  - CHRU Tours, Tours
  - CH Valence, Valence